CLINICAL TRIAL: NCT00941629
Title: Randomized Controlled Equivalence Trial Comparing Videoconference and Face-to-Face Delivery of Cognitive Processing Therapy for PTSD
Brief Title: Comparison of Videoconference and Face-to-Face Delivery of Cognitive Processing Therapy for Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSLC-IRB #H2013-0037; PT075415 (Other Grant/Funding Number: DOD PT075415)
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: PTSD; Telemedicine; Clinical Trial; Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Processing Therapy FTF (Active Comparator): Cognitive Processing Therapy delivered in traditional face-to-face sessions (FTF)
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)
- Cognitive Processing Therapy TMH (Experimental): Cognitive Processing Therapy delivered over videoconferencing equipment to a distant location (or telemental health; TMH)
  Interventions: Behavioral: Cognitive Processing Therapy (CPT)

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy (CPT) — Patients with PTSD receive a trauma-focused, cognitive-behavioral intervention in Face-to -Face treatment.
  Other Names: CPT
  Arms: Cognitive Processing Therapy FTF
Behavioral: Cognitive Processing Therapy (CPT) — Provision of Cognitive Processing Therapy over teleconference network (telemental health; telehealth)
  Other Names: CPT
  Arms: Cognitive Processing Therapy TMH

SUMMARY:
The purpose of this study is to evaluate the equivalence of CPT treatment delivered remotely via telemental health (TMH) over videoconferencing or via traditional face-to face (FTF) treatment to veterans who have Post-traumatic Stress Disorder (PTSD) from a military-related stressor (i.e., combat, sexual assault, non-combat physical assault). The secondary objective is to determine if patients' ratings of PTSD symptoms, affect, social adjustment, therapy alliance, treatment satisfaction and therapist satisfaction, are equivalent between service-delivery conditions (TMH vs. FTF). A final objective is to develop web-based practice assignments to assist participants in the TMH condition with treatment adherence (completion of the between- session practice assignments).

DETAILED DESCRIPTION:
PTSD is the most common mental health diagnosis affecting service men and women who have served in Iraq and Afghanistan (OEF/OIF). Despite unprecedented efforts by the Dept. of Defense (DoD) and Dept. of Veterans Affairs (VA) to treat these service personnel with mental disorders, significant gaps in the continuum of care for psychological health remain, specifically related to which services are offered, where services are offered, and who receives services. The DoD and VA have also attempted to address problems with accessibility through the development of a video teleconference (VTC) network to ensure that service members have access to top-quality specialized medical care regardless of their geographical location. Provision of medical treatment over VTC is often referred to as telemedicine; telemental health (TMH) refers to the provision of mental health treatment over the same system. A handful of studies have shown that psychiatry (primarily medication management) delivered over TMH systems can be as effective as face-to-face (FTF) treatment as long as the equipment and band-width are capable of delivering the communication in near real time.TMH is an increasingly common method of providing psychological treatment to service members with PTSD and other mental health problems, and yet there are no randomized trials of TMH provision of an empirically validated treatment for PTSD compared with FTF treatment. Therefore, this study aims to evaluate the treatment outcomes of patients with PTSD treated with CPT either remotely via TMH or traditionally in FTF treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Literate in written English
* Fluent in spoken English
* Verified status as an OEF/OIF veteran
* Current PTSD diagnosis
* Index traumatic event related to military services
* If taking psychotropic medication, remains stable

Exclusion Criteria:

* Under 18 years of age
* Not literate in written English
* Not fluent in spoke English
* Current uncontrolled psychotic or bipolar disorder
* Substance dependence
* Current uncontrolled suicidal or homicidal ideation
* Significant cognitive impairment that would interfere with completion of therapy tasks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The Clinician Administered PTSD Scale(CAPS) score. | At baseline, post-treatment( after 6 weeks) and the 3-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Tracey L Smith, Ph.D., Principal Investigator — Wm.S. Middleton Memorial Veterans Hospital FWA 00005784
Locations (2):
- United States (2):
  - Edward J. Hines Jr. Veterans Hospital, Cares Research Foundation FWA00001322, Hines, Illinois
  - Wm. S.Middleton Memorial Veterans Hospital, Madison, Wisconsin

REFERENCES:
- [Derived] Miles SR, Smith TL, Maieritsch KP, Ahearn EP. Fear of Losing Emotional Control Is Associated With Cognitive Processing Therapy Outcomes in U.S. Veterans of Afghanistan and Iraq. J Trauma Stress. 2015 Oct;28(5):475-9. doi: 10.1002/jts.22036. Epub 2015 Sep 23. PMID 26397721